CLINICAL TRIAL: NCT05591599
Title: Diagnostic Value of Calponin 2 in Identifying Tubal Pregnancies
Acronym: CNN2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 12/22/DD-BVMD
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-10

CONDITIONS: Tubal Pregnancy
Keywords: CALPONIN 2; CNN2; ectopic pregnancy; tubal pregnancy
MeSH Terms: conditions — Pregnancy, Tubal; Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Use blood test to measure serum calponin 2 level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Women diagnosed with tubal pregnancy
  Interventions: Diagnostic Test: calponin 2
- Control group: Women with the age corresponding to the case group (matched with the same age or +/- 2 years difference compared with the case group), diagnosed with spontaneous abortion or viable intrauterine pregnancy
  Interventions: Diagnostic Test: calponin 2

INTERVENTIONS:
Diagnostic Test: calponin 2 — serum calponin 2 level

SUMMARY:
Ectopic pregnancy (EP) is the implantation of a fertilized egg outside the main cavity of the uterus. EP is one of the most common gynecologic surgical emergencies , and one of leading causes of maternal mortality in the first trimester of pregnancy. Embryo implantation exerts different pressure on uterine and tubal epithelial and smooth muscle cells, calponin 2 (CNN2) expression at the implantation site would differ between intrauterine pregnancy and tubal pregnancy. The investigators conduct this study to find out the diagnostic value of CNN2 in identifying tubal pregnancies.

DETAILED DESCRIPTION:
This is a case-control prospective study. Women age 18-35 years old, come to My Duc, My Duc phu Nhuan Hospital and Ngoc Lan Clinic and have the indication of testing beta human chorionic gonadotropin (hCG) for determining pregnancy status because of 1-14 days period delay with or without abdominal pain, vaginal bleeding or after assisted reproductive technology. Those women will be introduced about the study. If they agree to take part in and write the consent form, they will be taken 5ml of blood more at the same time of testing beta hCG. Blood sample will then be centrifuged and collected serum will then be stored at -80 celsius degree.

Women with negative beta hCG will be excluded. Women with positive beta hCG will be followed-up pregnancy as routine until 12 6/7 weeks of gestational age (GA). At this time, those women will be screened using including and excluding criteria for each group. They then be put group into (1) tubal pregnancy, (2) viable pregnancy and (3) early pregnancy loss.

Stored serum sample will be defrosted and measured CNN2 concentration.

ELIGIBILITY:
Case: tubal pregnancy

* Inclusion criteria

  * Patients aged 18 years to < 35 years old
  * Positive beta-hCG result
  * Diagnosed with tubal pregnancy based on pathological result.
* Exclusion criteria

  * BMI > 30 kg/m2
  * A co-existing additional pregnancy
  * Refuse to participate in the study

Control group: Women with the age corresponding to the case group (matched with the same age or +/- 2 years difference compared with the case group), diagnosed with early pregnancy loss or viable intrauterine pregnancy.

Early pregnancy loss

* Inclusion criteria

  * Patients aged 18 years old to < 35 years old
  * Positive beta-hCG result
  * Pregnancy outcome recorded as early pregnancy loss: ultrasound shows an empty gestational sac in the uterus or a gestational sac with embryos but no fetal cardiac activity within the first 12 weeks 6/7 days of pregnancy. Or there is pathological pathology of the specimen taken from the uterine lumen as placenta or fetal tissue.
* Exclusion criteria

  * BMI > 30 kg/m2
  * A co-existing ectopic pregnancy
  * Refuse to participate in the study

Viable intrauterine pregnancy

* Inclusion criteria

  * Patients aged 18 years old to < 35 years old
  * Transvaginal ultrasound records images of a living fetus in the uterine with embryos and fetal heart activity until 12 6/7 weeks of gestation (ultrasound or last menstrual period)
* Exclusion criteria

  * BMI > 30 kg/m2
  * A co-existing ectopic pregnancy
  * Multiple pregnancies
  * Refuse to participate in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to <35 years old, coming to the clinic because their period is 1-14 days delay with or without abdominal pain, vaginal bleeding, or women at this age come to the clinic for follow-up after assisted reproductive technology at Ngoc Lan clinic, My Duc hospital, My Duc Phu Nhuan; and had a positive beta-hCG result.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The average serum CNN2 level | Up to 12 6/7 weeks of gestational age
  The average serum CNN2 level of each group

SECONDARY OUTCOMES:
The average beta hCG level | Up to 12 6/7 weeks of gestational age
  The average beta hCG level of each group

CONTACTS AND LOCATIONS:
Overall Officials: Minh N Chau, MD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barnhart KT. Clinical practice. Ectopic pregnancy. N Engl J Med. 2009 Jul 23;361(4):379-87. doi: 10.1056/NEJMcp0810384. No abstract available. PMID 19625718
- [Result] Shaw JL, Dey SK, Critchley HO, Horne AW. Current knowledge of the aetiology of human tubal ectopic pregnancy. Hum Reprod Update. 2010 Jul-Aug;16(4):432-44. doi: 10.1093/humupd/dmp057. Epub 2010 Jan 12. PMID 20071358
- [Result] Senapati S, Barnhart KT. Biomarkers for ectopic pregnancy and pregnancy of unknown location. Fertil Steril. 2013 Mar 15;99(4):1107-16. doi: 10.1016/j.fertnstert.2012.11.038. Epub 2013 Jan 3. PMID 23290746
- [Result] Bobdiwala S, Al-Memar M, Farren J, Bourne T. Factors to consider in pregnancy of unknown location. Womens Health (Lond). 2017 Aug;13(2):27-33. doi: 10.1177/1745505717709677. Epub 2017 Jun 29. PMID 28660799
- [Result] Wang DJ, Huang H, Wang HY, Yuan H, Du P, Wang CY, Wang YF. Association study of vascular endothelial growth factor gene polymorphisms with ectopic pregnancy in Chinese women. Clin Exp Obstet Gynecol. 2014;41(6):665-70. PMID 25551960
- [Result] Felemban A, Sammour A, Tulandi T. Serum vascular endothelial growth factor as a possible marker for early ectopic pregnancy. Hum Reprod. 2002 Feb;17(2):490-2. doi: 10.1093/humrep/17.2.490. PMID 11821301
- [Result] Rausch ME, Barnhart KT. Serum biomarkers for detecting ectopic pregnancy. Clin Obstet Gynecol. 2012 Jun;55(2):418-23. doi: 10.1097/GRF.0b013e31825109f6. PMID 22510623
- [Result] Mueller MD, Raio L, Spoerri S, Ghezzi F, Dreher E, Bersinger NA. Novel placental and nonplacental serum markers in ectopic versus normal intrauterine pregnancy. Fertil Steril. 2004 Apr;81(4):1106-11. doi: 10.1016/j.fertnstert.2003.08.049. PMID 15066471
- [Result] Senapati S, Sammel MD, Butts SF, Takacs P, Chung K, Barnhart KT. Predicting first trimester pregnancy outcome: derivation of a multiple marker test. Fertil Steril. 2016 Dec;106(7):1725-1732.e3. doi: 10.1016/j.fertnstert.2016.08.044. Epub 2016 Oct 26. PMID 28340932
- [Result] Rausch ME, Sammel MD, Takacs P, Chung K, Shaunik A, Barnhart KT. Development of a multiple marker test for ectopic pregnancy. Obstet Gynecol. 2011 Mar;117(3):573-582. doi: 10.1097/AOG.0b013e31820b3c61. PMID 21343760
- [Result] Wijayarathna R, de Kretser DM. Activins in reproductive biology and beyond. Hum Reprod Update. 2016 Apr;22(3):342-57. doi: 10.1093/humupd/dmv058. Epub 2016 Feb 15. PMID 26884470
- [Result] Florio P, Severi FM, Bocchi C, Luisi S, Mazzini M, Danero S, Torricelli M, Petraglia F. Single serum activin a testing to predict ectopic pregnancy. J Clin Endocrinol Metab. 2007 May;92(5):1748-53. doi: 10.1210/jc.2006-2188. Epub 2007 Mar 6. PMID 17341564
- [Result] Zhao Z, Zhao Q, Warrick J, Lockwood CM, Woodworth A, Moley KH, Gronowski AM. Circulating microRNA miR-323-3p as a biomarker of ectopic pregnancy. Clin Chem. 2012 May;58(5):896-905. doi: 10.1373/clinchem.2011.179283. Epub 2012 Mar 6. PMID 22395025
- [Result] Zhang R, Li S, Wang Y, Cai W, Liu Q, Zhang J. Serum calponin 2 is a novel biomarker of tubal ectopic pregnancy. Fertil Steril. 2021 Oct;116(4):1020-1027. doi: 10.1016/j.fertnstert.2021.05.101. Epub 2021 Jul 1. PMID 34217487
- [Result] Liu R, Jin JP. Calponin isoforms CNN1, CNN2 and CNN3: Regulators for actin cytoskeleton functions in smooth muscle and non-muscle cells. Gene. 2016 Jul 1;585(1):143-153. doi: 10.1016/j.gene.2016.02.040. Epub 2016 Mar 10. PMID 26970176
- [Result] Hossain MM, Crish JF, Eckert RL, Lin JJ, Jin JP. h2-Calponin is regulated by mechanical tension and modifies the function of actin cytoskeleton. J Biol Chem. 2005 Dec 23;280(51):42442-53. doi: 10.1074/jbc.M509952200. Epub 2005 Oct 18. PMID 16236705